CLINICAL TRIAL: NCT07368582
Title: Real World Pediatric Oncology Rehabilitation in Italy (ReWori) Study Protocol: Prognostic Factors of Functional Abilities in Children, Adolescents and Young Adults With Cancer Undergoing Rehabilitation
Brief Title: Real World Pediatric Oncology Rehabilitation in Italy ( ReWori )
Acronym: REWORI
Status: Recruiting | Type: Observational
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Sponsor
Other Study IDs: REWORI; AIEOP (Other: AIEOP - Associazione Italiana Ematologia Oncologia Pediatrica)
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Pediatric Cancer Patients; Pediatric Oncology; Rehabilitation; Motor Outcomes; Physical Therapy
Keywords: pediatric oncology; rehabilitation; motor performance; physical therapy; children; adolescents; young adults; exercise
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitation intervention — This is an observational study, so it does not have a specific rehabilitation treatment protocol to be followed. The chort is followed with a periodic evaluation (monthly or every three month only for bone tumour diagnosis) during the period of the rehabilitation treatment

SUMMARY:
This observational study aims to describe changes in the functional abilities of children, adolescents and young adults with cancer who are undergoing physiotherapy or neuropsychomotor rehabilitation. This is real-world study aiming to describe normal rehabilitation pathways in many different hospitals or rehabilitation centres in Italy.

The primary research question is:

1) What are the longitudinal changes in functional abilities among these patients receiving physiotherapy or neuropsychomotor rehabilitation?

The secondary research questions are:

1. What types of rehabilitation practices are implemented across AIEOP centres?
2. What are the rehabilitation needs among patients undergoing physiotherapy or neuropsychomotor rehabilitation?
3. How does health-related quality of life differ across the various stages of the rehabilitation pathway? Participants undergoing usual rehabilitation treatment are evaluated on their functional abilities on a monthly basis. If they agree to participate in this study, the main characteristics of the rehabilitation treatment and the monthly evaluation are collected.

DETAILED DESCRIPTION:
Each year in Italy, about 1,400 children, 800 adolescents are diagnosed with cancer, with survival rates approaching 80percent. Despite improved survival, cancer and its treatments often lead to functional impairments and delays in neuropsychomotor development, affecting the musculoskeletal, nervous, and cardiovascular systems. These limitations can occur throughout all phases of care, from diagnosis to post-treatment, making rehabilitation increasingly important to preserve and improve quality of life. Although rehabilitation is recognized as beneficial in paediatric oncology, current evidence on the effectiveness of physiotherapy and neuropsychomotor interventions remains limited. Research has largely focused on general physical activity rather than targeted rehabilitation aimed at restoring specific functions such as mobility, balance, or joint function. A 2021 Cochrane review highlighted the need for high-quality, multicentre studies with standardized protocols, homogeneous patient groups, clearly defined and measurable outcomes, and long-term follow-up.

Currently, there are no shared international guidelines or Core Outcome Sets (COS) for rehabilitation in paediatric oncology. To address this gap, the Italian Association of Paediatric Haematology and Oncology (AIEOP) developed consensus-based recommendations for rehabilitation assessment and treatment and promoted the validation of the Functional Abilities Assessment in Paediatric Oncology (FAAP-O) scale. However, there is still the lack of data on prognostic factors influencing functional outcomes, rehabilitation needs, and types of rehabilitation care provided to children, adolescents, and young adults with cancer.

The primary objective is to describe changes in functional abilities in patients undergoing physiotherapy or neuropsychomotor rehabilitation. Secondary objectives include describing rehabilitation practices across AIEOP centres, estimating rehabilitation needs, and assessing quality of life at different stages of rehabilitation. The main endpoint is represented by functional ability levels, which are measured using the FAAP-O scale for patients with all types of cancer except bone tumours, and the TESS-pTESS questionnaires for patients with bone tumours. Secondary endpoints include rehabilitation tools, rehabilitation goals, treatment intensity, types of exercises, incidence of rehabilitation referrals with related impairments, and quality of life measured using the PedsQL and Bt-DUX questionnaires. The study will be conducted in compliance with Good Clinical Practice guidelines and the Declaration of Helsinki. Ethical approval from local ethics committees is required before patient enrolment, and no external funding is provided for the study. Patient confidentiality will be ensured through anonymised data collection. Each participant will be assigned a centre specific alphanumeric code. Personal identifiers will be accessible only to the enrolling centre. The year of birth will be recorded to minimize data entry errors.

All participants, or their legal guardians, will receive detailed information about the study objectives, data handling, and confidentiality measures. Participation is voluntary and will not affect rehabilitation care. Written informed consent will be obtained prior to enrolment. Data analysis will include descriptive statistics for continuous and categorical variables. Changes in functional abilities over time will be evaluated using paired statistical tests, while mixed-effects regression models will be used to explore associations between predictors and outcomes in a multicentre, longitudinal framework. Statistical significance will be set at 5%. Based on the primary outcome measures (FAAP-O, pTESS, and TESS), a sample size of 199 participants is required to detect a small effect size (0.20) with 80% power. Accounting for an anticipated 20% dropout rate, the total enrolment target is 249 patients. A rehabilitation assessment will be carried out upon referral to the rehabilitation service and then on a monthly basis throughout the rehabilitation process. Data will be collected electronically using an online case report form (CRF) on the REDCap platform, accessible to all participating centres following the ethical committee approbation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer,
* Children, adolescents and young adults aged between 0 and 24 years old,
* Children, adolescents and young adults at any stage of treatment and off therapy,
* Children, adolescents and young adults referred to the Rehabilitation Service of AIEOP centres and Rehabilitation Centres that provide rehabilitation care for paediatric and young adult cancer patients involved in the study.

Exclusion Criteria:

* Failure to sign the consent/assent form for participation in the study by the subject and/or by the person exercising parental authority.

Ages: 0 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults aged between 0 and 24 years old with a diagnosis of cancer at any stage of treatment and off therapy. They must be referred to the Rehabilitation Service of AIEOP centres and Rehabilitation Centres that provide rehabilitation care for paediatric and young adult cancer patients involved in the study
Sampling Method: Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Functional Abilities Assessment in Pediatric Oncology (FAAP-O) | One month
  The Functional Abilities Assessment in Pediatric Oncology (FAAP-O) scale assesses global motor abilities in children and adolescents with cancer through 36 items. Scores range from 0 to 3, where 0 indicates that the child does not initiate the task, 1 initiates the task (<10%), 2 partially completes the task (10% to <100%), and 3 completes the task as described in the criteria. Higher scores mean a better outcome. It is validated for children and adolescents aged 6 months to 18 years.
Toronto Extremity Salvage Score (TESS) | Three months
  The Toronto ExtremitySalvage Score (TESS) isa self-administered questionnaire used to assess subjective functional abilities and residual disability in patients with musculoskeletal oncological diseases. Through30 items, patients are asked to rate perceived difficulty in performing specific activities. The tasks are rated from 0 (not possible) to 5 (without any problem). The raw score is converted to a score ranging from 0 to 100 points, with higher scores indicating a less functional limitation. It can be administered from the age of 12 years.
Pediatric Toronto Extremity Salvage Score (pTESS) | Three months
  The Pediatric Toronto ExtremitySalvage Score (pTESS) is self-administered questionnaire. Is the pediatric version of the TESS, adapted and validated for children and adolescents with bone tumors. The Ptess comprehends 30 items. Each item is an swered using a 5-point ordinal scale, and all item responses are aggregated into a single summary score. Five points are allotted for the first response option ("not at all hard"), 4 points for the second option, and so on, until 1 point is allotted for the fifth option("too hard. I can't"). Each item has a "not applicable" option, phrased as: "I do not do this." This not applicable (NA) option is notgiven a numeric score and for scoring is considered invalid. Summary scores indicate physical function ranging from 0 (lowest) to 100 (highest).It can be used from the age of 7 years.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory™ (PedsQL) | One month
  The PedsQL questionnaire measures health-related quality of life in children and young people. There are two versions: a parent proxy version and a children's version. These are divided in differentage ranges (subjects aged 2-4 years, 5-7 years, 8-12 years, 13-18 years and 18-25 years). PedsQL includes 23 items across four domains: physical, emotional, social, and school functioning. The scoring system is based on a 5-point Likert scale (0-4), where 0 means "Never a problem" and 4 means "Almost always a problem" that is reversed-scored and transformed to a 0-100 scale, where higher scores indicate better health-related quality of life (0=100, 1=75, 2=50, 3=25, 4=0). It calculates scores by averaging items within subscales (physical, emotional, social, school). It is validated from 2 to18 years old.
DUX for Bone Tumors in Children and Adolescents (Bt-DUX) | Three months
  The Bt-DUX questionnaire identifies health-related quality of life in patients who have undergone surgery for malignant bone tumors of the lower limb. It consists of 20 items addressing social, emotional, aesthetic, and physical aspects. Each item can be scored using a five-point Likert scale ranging from 1, which means "very happy", to 5, which means "sad". These single-item scores are then converted in to total and domain scores. These raw scores are then converted into total and domain scores ranging from 0 to 100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Rossi Rossi, Master's degree, Principal Investigator — AOU Città della Salute e della Scienza di Torino - Ospedale Infantile Regina Margherita
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy